CLINICAL TRIAL: NCT03294031
Title: Pilates as an Adjuvant Physical Exercise Therapy in Patients With Parkinson Disease.
Brief Title: Pilates as an Adjuvant Therapy in Parkinson Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Gustavo Rodríguez Fuentes, Ph.D., University of Vigo
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015/484
Record Dates: First submitted 2017-09-18; First posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Neurodegenerative Disorder; Physical Activity; Pilates Method; Stabilometer
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases; Motor Activity | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates (Experimental): The Pilates program covered a 12-week period, two weekly sessions. In one session, exercises were performed on a mat (Mat Pilates), and in the second session in standing and sitting position. The programme included warm-up exercises, the main part of the session and cooling activities.
  Interventions: Other: Pilates
- Conventional Exercise (Active Comparator): The conventional exercise programme covered a 12-week period, two weekly sessions. The programme aimed at improving aerobic capacity, muscular resistance, balance and flexibility. The program combined land-based and water-based exercise sessions.
  Interventions: Other: Conventional Exercise

INTERVENTIONS:
Other: Pilates — Warm-up exercises included Abdominal and costal breathing and Pelvic Clock. Some exercises included in the main part of the mat session were Arm arcs, Curls up, Femur arcs, Shoulder bridge, Leg circles, among others. The main part of the sitting/standing session included in standing position exercises like Standing on one leg with support, Neck rolls, Side leg lift with support and in sitting position Spine stretch 5", Elbows back with hands behind his head, Heel/knee slides, Shoulder drops, Knee folds, among others. In mat sessions, cooling exercises included in standing position Hamstring stretch and Abdominal Breathing and Rest position and in sitting/standing session Stretching and Abdominal Breathing.
  Arms: Pilates
Other: Conventional Exercise — All sessions started with a 15-minute warm-up phase based on walking performance and joint mobility exercises. It was followed by a 35-minute second phase, which included low-impact aerobics (music tempo was set at 120 beats per minute), gross motor coordination tasks and balance activities. The final 5-minute phase focused on gentle stretching exercises.
  Arms: Conventional Exercise

SUMMARY:
Although Pilates has been proposed as a useful rehabilitation strategy in PD, research on its feasibility and potential effects on the motor symptoms and balance with this population is scarce. Some works have included Pilates as part of combined exercise session interventions, but information concerning their specific effects was not provided. Under these circumstances, this study aims at identifying the effects of adding Pilates as part of a conventional exercise rehabilitation program on the motor symptoms and static balance of PD persons. Participants (n=15) were assigned to a Pilates (PG) or to a conventional exercise group (CG) and performed one land-based and one water-based exercise session per week for 14 weeks. The MDS-UPDRS and a stabilometer were used to assess the impact of the intervention on the participant´s motor symptoms and static balance.

ELIGIBILITY:
Inclusion Criteria:

* Stages 1 through 3 on the Hoehn and Yahr Staging Scale;
* Stable reaction to anti-Parkinson medication;
* Not having taken part in any physical exercise program during the month prior to the study.

Exclusion Criteria:

* People with PD who were not able to ambulate independently or presented any comorbidities other than PD or any acute illness that would make training inappropriate.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2016-05-27 (Actual); Study Completion 2016-05-27 (Actual)

PRIMARY OUTCOMES:
Motor impairment. | The participants were assessed one week before starting the program (week #0).
  The Spanish adapted version of the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) was administered to assess the impact of the intervention on the motor impairment and disability related to PD. The MDS-UPDRS total score ranges from zero to 200, with higher scores indicating a greater impact of PD symptoms.

SECONDARY OUTCOMES:
Anthropometric Measurements. | The participants were assessed one week before starting the program (week #0).
  The height (cm) and weight (kg) of the participants were measured without shoes and in light clothing. The body mass index (BMI) was calculated using the following formula: weight / height2 (kg/m2).
Change from baseline Anthropometric Measurements at week 15. | The participants were assessed one week after the programme was completed (week #15).
  The height (cm) and weight (kg) of the participants were measured without shoes and in light clothing. The body mass index (BMI) was calculated using the following formula: weight / height2 (kg/m2).
Change from week 15 Anthropometric Measurements at week 18 follow-up. | Follow-up assessment was performed four weeks after training ended (week #18).
  The height (cm) and weight (kg) of the participants were measured without shoes and in light clothing. The body mass index (BMI) was calculated using the following formula: weight / height2 (kg/m2).
Static Balance at baseline. | The participants were assessed one week before starting the program (week #0).
  The static balance was evaluated using the TecnoBody Prokin 3 platform. The assessment protocol was developed in a sitting and standing position, with open (OE) and closed (CE) eyes. The participants had three 30-second attempts to perform the position with open and closed eyes and a 60-second interval of active rest between them. The static balance parameters assessed were the centre of pressure of the body in the frontal plane, the centre of pressure of the body in the sagittal plane, the amplitude movement of the centre of pressure in the sagittal plane, the amplitude movement of the centre of pressure in the frontal plane, the average speed of oscillation movement of the centre of pressure in the sagittal plane, the average speed of oscillation movement of the centre of pressure in the frontal plane, the sum of distances of the amount of movement of the centre of pressure, and the displacement area of the centre of pressure.
Change from baseline Static Balance at 15 weeks. | The participants were assessed one week after the programme was completed (week #15).
  The static balance was evaluated using the TecnoBody Prokin 3 platform. The assessment protocol was developed in a sitting and standing position, with open (OE) and closed (CE) eyes. The participants had three 30-second attempts to perform the position with open and closed eyes and a 60-second interval of active rest between them. The static balance parameters assessed were the centre of pressure of the body in the frontal plane, the centre of pressure of the body in the sagittal plane, the amplitude movement of the centre of pressure in the sagittal plane, the amplitude movement of the centre of pressure in the frontal plane, the average speed of oscillation movement of the centre of pressure in the sagittal plane, the average speed of oscillation movement of the centre of pressure in the frontal plane, the sum of distances of the amount of movement of the centre of pressure, and the displacement area of the centre of pressure.
Change from week 15 Static Balance at week 18 follow-up. | Follow-up assessment was performed four weeks after training ended (week #18).
  The static balance was evaluated using the TecnoBody Prokin 3 platform. The assessment protocol was developed in a sitting and standing position, with open (OE) and closed (CE) eyes. The participants had three 30-second attempts to perform the position with open and closed eyes and a 60-second interval of active rest between them. The static balance parameters assessed were the centre of pressure of the body in the frontal plane, the centre of pressure of the body in the sagittal plane, the amplitude movement of the centre of pressure in the sagittal plane, the amplitude movement of the centre of pressure in the frontal plane, the average speed of oscillation movement of the centre of pressure in the sagittal plane, the average speed of oscillation movement of the centre of pressure in the frontal plane, the sum of distances of the amount of movement of the centre of pressure, and the displacement area of the centre of pressure.
Change from baseline Motor Impairment at 15 weeks. | The participants were assessed one week after the programme was completed (week #15).
  The Spanish adapted version of the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) was administered to assess the impact of the intervention on the motor impairment and disability related to PD. The MDS-UPDRS total score ranges from zero to 200, with higher scores indicating a greater impact of PD symptoms.
Change from week 15 Motor Impairment at week 18 follow-up. | Follow-up assessment was performed four weeks after training ended (week #18).
  The Spanish adapted version of the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) was administered to assess the impact of the intervention on the motor impairment and disability related to PD. The MDS-UPDRS total score ranges from zero to 200, with higher scores indicating a greater impact of PD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: José María Cancela-Carral, Ph.D., Study Director — University of Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbruzzese G, Marchese R, Avanzino L, Pelosin E. Rehabilitation for Parkinson's disease: Current outlook and future challenges. Parkinsonism Relat Disord. 2016 Jan;22 Suppl 1:S60-4. doi: 10.1016/j.parkreldis.2015.09.005. Epub 2015 Sep 3. PMID 26360239
- [Background] Ayan C, Cancela JM, Gutierrez-Santiago A, Prieto I. Effects of two different exercise programs on gait parameters in individuals with Parkinson's disease: a pilot study. Gait Posture. 2014;39(1):648-51. doi: 10.1016/j.gaitpost.2013.08.019. Epub 2013 Sep 7. PMID 24021522
- [Background] Di Giulio I, St George RJ, Kalliolia E, Peters AL, Limousin P, Day BL. Maintaining balance against force perturbations: impaired mechanisms unresponsive to levodopa in Parkinson's disease. J Neurophysiol. 2016 Aug 1;116(2):493-502. doi: 10.1152/jn.00996.2015. Epub 2016 Apr 20. PMID 27098030
- [Background] Dibble LE, Addison O, Papa E. The effects of exercise on balance in persons with Parkinson's disease: a systematic review across the disability spectrum. J Neurol Phys Ther. 2009 Mar;33(1):14-26. doi: 10.1097/NPT.0b013e3181990fcc. PMID 19265767
- [Background] Johnson L, Putrino D, James I, Rodrigues J, Stell R, Thickbroom G, Mastaglia FL. The effects of a supervised Pilates training program on balance in Parkinson's disease. Advances in Parkinson Disease 2: 58-61, 2013.
- [Background] Kalron A, Rosenblum U, Frid L, Achiron A. Pilates exercise training vs. physical therapy for improving walking and balance in people with multiple sclerosis: a randomized controlled trial. Clin Rehabil. 2017 Mar;31(3):319-328. doi: 10.1177/0269215516637202. Epub 2016 Jul 10. PMID 26951348
- [Background] Kamioka H, Tsutani K, Katsumata Y, Yoshizaki T, Okuizumi H, Okada S, Park SJ, Kitayuguchi J, Abe T, Mutoh Y. Effectiveness of Pilates exercise: A quality evaluation and summary of systematic reviews based on randomized controlled trials. Complement Ther Med. 2016 Apr;25:1-19. doi: 10.1016/j.ctim.2015.12.018. Epub 2016 Jan 4. PMID 27062942
- [Background] King LA, Horak FB. Delaying mobility disability in people with Parkinson disease using a sensorimotor agility exercise program. Phys Ther. 2009 Apr;89(4):384-93. doi: 10.2522/ptj.20080214. Epub 2009 Feb 19. PMID 19228832
- [Background] Klamroth S, Steib S, Devan S, Pfeifer K. Effects of Exercise Therapy on Postural Instability in Parkinson Disease: A Meta-analysis. J Neurol Phys Ther. 2016 Jan;40(1):3-14. doi: 10.1097/NPT.0000000000000117. PMID 26655098
- [Background] Martinez-Martin P, Rodriguez-Blazquez C, Alvarez-Sanchez M, Arakaki T, Bergareche-Yarza A, Chade A, Garretto N, Gershanik O, Kurtis MM, Martinez-Castrillo JC, Mendoza-Rodriguez A, Moore HP, Rodriguez-Violante M, Singer C, Tilley BC, Huang J, Stebbins GT, Goetz CG. Expanded and independent validation of the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS). J Neurol. 2013 Jan;260(1):228-36. doi: 10.1007/s00415-012-6624-1. Epub 2012 Aug 5. PMID 22865238
- [Background] Santamato A, Ranieri M, Panza F, Zoccolella S, Frisardi V, Solfrizzi V, Amoruso MT, Amoruso L, Fiore P. Botulinum toxin type A and a rehabilitation program in the treatment of Pisa syndrome in Parkinson's disease. J Neurol. 2010 Jan;257(1):139-41. doi: 10.1007/s00415-009-5310-4. No abstract available. PMID 19763384
- [Result] Ayan C, Varela S, Vila MH, Seijo-Martinez M, Cancela JM. Treadmill training combined with water and land-based exercise programs: Effects on Parkinson's disease patients. NeuroRehabilitation. 2016 Jun 30;39(2):295-9. doi: 10.3233/NRE-161360. PMID 27372364
- [Result] Bergamin M, Gobbo S, Bullo V, Zanotto T, Vendramin B, Duregon F, Cugusi L, Camozzi V, Zaccaria M, Neunhaeuserer D, Ermolao A. Effects of a Pilates exercise program on muscle strength, postural control and body composition: results from a pilot study in a group of post-menopausal women. Age (Dordr). 2015 Dec;37(6):118. doi: 10.1007/s11357-015-9852-3. Epub 2015 Nov 15. PMID 26578458
- [Result] Bird ML, Hill KD, Fell JW. A randomized controlled study investigating static and dynamic balance in older adults after training with Pilates. Arch Phys Med Rehabil. 2012 Jan;93(1):43-9. doi: 10.1016/j.apmr.2011.08.005. Epub 2011 Oct 5. PMID 21975148
- [Result] Cattaneo D, Jonsdottir J, Regola A, Carabalona R. Stabilometric assessment of context dependent balance recovery in persons with multiple sclerosis: a randomized controlled study. J Neuroeng Rehabil. 2014 Jun 10;11:100. doi: 10.1186/1743-0003-11-100. PMID 24912561
- [Result] Bang DH, Cho HS. Effect of body awareness training on balance and walking ability in chronic stroke patients: a randomized controlled trial. J Phys Ther Sci. 2016 Jan;28(1):198-201. doi: 10.1589/jpts.2016.198. Epub 2016 Jan 30. PMID 26957757
- [Result] de Oliveira Francisco C, de Almeida Fagundes A, Gorges B. Effects of Pilates method in elderly people: Systematic review of randomized controlled trials. J Bodyw Mov Ther. 2015 Jul;19(3):500-8. doi: 10.1016/j.jbmt.2015.03.003. Epub 2015 Mar 20. PMID 26118523
- [Result] Donath L, Roth R, Hurlimann C, Zahner L, Faude O. Pilates vs. Balance Training in Health Community-Dwelling Seniors: a 3-arm, Randomized Controlled Trial. Int J Sports Med. 2016 Mar;37(3):202-10. doi: 10.1055/s-0035-1559695. Epub 2015 Dec 2. PMID 26630547
- [Result] Guclu-Gunduz A, Citaker S, Irkec C, Nazliel B, Batur-Caglayan HZ. The effects of pilates on balance, mobility and strength in patients with multiple sclerosis. NeuroRehabilitation. 2014;34(2):337-42. doi: 10.3233/NRE-130957. PMID 23949064
- [Result] King LA, Salarian A, Mancini M, Priest KC, Nutt J, Serdar A, Wilhelm J, Schlimgen J, Smith M, Horak FB. Exploring outcome measures for exercise intervention in people with Parkinson's disease. Parkinsons Dis. 2013;2013:572134. doi: 10.1155/2013/572134. Epub 2013 Apr 30. PMID 23738230
- [Result] Kucuk F, Kara B, Poyraz EC, Idiman E. Improvements in cognition, quality of life, and physical performance with clinical Pilates in multiple sclerosis: a randomized controlled trial. J Phys Ther Sci. 2016 Mar;28(3):761-8. doi: 10.1589/jpts.28.761. Epub 2016 Mar 31. PMID 27134355
- [Result] La Touche R, Escalante K, Linares MT. Treating non-specific chronic low back pain through the Pilates Method. J Bodyw Mov Ther. 2008 Oct;12(4):364-70. doi: 10.1016/j.jbmt.2007.11.004. Epub 2008 Feb 1. PMID 19083695
- [Result] Lange C, Unnithan VB, Larkam E, Latta PM. Maximizing the benefits of Pilates-inspired exercise for learning functional motor skills. Journal of Bodywork and Movement Therapies 4: 99-108, 2000.
- [Result] Markovic G, Sarabon N, Greblo Z, Krizanic V. Effects of feedback-based balance and core resistance training vs. Pilates training on balance and muscle function in older women: a randomized-controlled trial. Arch Gerontol Geriatr. 2015 Sep-Oct;61(2):117-23. doi: 10.1016/j.archger.2015.05.009. Epub 2015 May 27. PMID 26036209
- [Result] Phrompaet S, Paungmali A, Pirunsan U, Sitilertpisan P. Effects of pilates training on lumbo-pelvic stability and flexibility. Asian J Sports Med. 2011 Mar;2(1):16-22. doi: 10.5812/asjsm.34822. PMID 22375213
- [Result] Schmitz-Hubsch T, Pyfer D, Kielwein K, Fimmers R, Klockgether T, Wullner U. Qigong exercise for the symptoms of Parkinson's disease: a randomized, controlled pilot study. Mov Disord. 2006 Apr;21(4):543-8. doi: 10.1002/mds.20705. PMID 16229022
- [Result] Tolnai N, Szabo Z, Koteles F, Szabo A. Physical and psychological benefits of once-a-week Pilates exercises in young sedentary women: A 10-week longitudinal study. Physiol Behav. 2016 Sep 1;163:211-218. doi: 10.1016/j.physbeh.2016.05.025. Epub 2016 May 16. PMID 27195456
- [Result] Volpe D, Giantin MG, Maestri R, Frazzitta G. Comparing the effects of hydrotherapy and land-based therapy on balance in patients with Parkinson's disease: a randomized controlled pilot study. Clin Rehabil. 2014 Dec;28(12):1210-7. doi: 10.1177/0269215514536060. Epub 2014 Jun 3. PMID 24895382
- [Result] Wells C, Kolt GS, Marshall P, Bialocerkowski A. Indications, benefits, and risks of Pilates exercise for people with chronic low back pain: a Delphi survey of Pilates-trained physical therapists. Phys Ther. 2014 Jun;94(6):806-17. doi: 10.2522/ptj.20130568. Epub 2014 Apr 3. PMID 24700138
- [Result] Wong-Yu IS, Mak MK. Multi-dimensional balance training programme improves balance and gait performance in people with Parkinson's disease: A pragmatic randomized controlled trial with 12-month follow-up. Parkinsonism Relat Disord. 2015 Jun;21(6):615-21. doi: 10.1016/j.parkreldis.2015.03.022. Epub 2015 Mar 31. PMID 25899544